CLINICAL TRIAL: NCT03341702
Title: Predictive Factors of Violence in Prison, Retrospective Study in an French Incarcerated Male Population
Brief Title: Predictive Factors of Violence in Prison
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0324
Record Dates: First submitted 2017-10-10; First posted 2017-11-14 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2017-10

CONDITIONS: Prisoner
Keywords: jail; violence; predictive factors; prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: penintetiary's incident reports collection — collection of clinical and penitentiary 's data

SUMMARY:
Prison concentrates people with violent behavior and patients suffering from psychiatric disorders. Aggression are daily, the suicide rate is 5 to 10 times higher than the ordinary environment and current prevention devices have shown their limits.

That's why, in order to improve the violence's prevention in prison, the investigator propose to identify the predictive factors of violence by studying retrospectively the link between the psychiatric profile and commission of violence after being jailed.

DETAILED DESCRIPTION:
From the 1st January to the 31 December 2012, every man incarcerated was screened thanks to the Mini International Neuropsychiatric Interview (MINI) to establish the presence of a current and/or past psychiatric diagnoses. In addition, collection of violent incidents based on penitentiary's reports (aggression, suicide, self-mutilation, intoxication, murder…) was conducted .

Then statistic analysis compared psychiatric characteristics of prisoners according to whether they commit violence or not within 12 months after being jailed, distinguish the authors of self and hetero aggressive violence. Those tests are completed with a cluster analysis to precise psychiatric from criminological profiles of dangerousness.

ELIGIBILITY:
Inclusion criteria:

- being jailed from 1st january 2012 to 31 dec 2012 in the Villeneuve Lès Maguelonne prison (Hérault, France)

Exclusion criteria:

- opposition form, unable to understand french, age under 18

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male incarcerated in a french prison
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
violent event | within the 12 month after incarceration
  physical assault
violent event | within the 12 month after incarceration
  suicide attempt
violent event | within the 12 month after incarceration
  intoxication
violent event | within the 12 month after incarceration
  violent death
violent event | within the 12 month after incarceration
  sexual assault
violent event | within the 12 month after incarceration
  fire

SECONDARY OUTCOMES:
suicide attempt | within the 12 month after incarceration
  according to the prison suicide attempt recording
physical assault | within the 12 month after incarceration
  according to the prison suicide attempt recording

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu LACAMBRE, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC